CLINICAL TRIAL: NCT02606617
Title: What is the Effects of Prokinetic Drug on the Blood Glucose in Type 2 Diabetes Patients: Mosapride Comparing Placebo
Brief Title: A Clinical Trial Analyzing Effects of Prokinetic Drug on the Blood Glucose in Patients With Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Zhiming Zhu, MD, PhD, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PDBG
Record Dates: First submitted 2015-10-25; First posted 2015-11-17 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Type 2 Diabetes
Keywords: Mosapride; blood glucose; serum lipid
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — mosapride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Mosapride (Active Comparator): Mosapride(5mg, 3/d), antidiabetic drug except DPP-IV inhibitor and GLP-1 receptor activator.
  Interventions: Drug: Mosapride
- Placebo (Placebo Comparator): Placebo(5mg, 3/d), antidiabetic drug except DPP-IV inhibitor and GLP-1 receptor activator.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mosapride — Mosapride(5mg, 3/d), antidiabetic drug except DPP-IV inhibitor and GLP-1 receptor activator.
  Arms: Mosapride
Drug: Placebo — Placebo(5mg, 3/d), antidiabetic drug except DPP-IV inhibitor and GLP-1 receptor activator.
  Arms: Placebo

SUMMARY:
With the improvement of living level, the incidence rates of diabetes, obesity, and hypertension in China increased quickly, which are 11.6%, 7.1% and 18.8% respectively, according to the newly investigated data. The clustering of diabetes, obesity, hypertension and dyslipidemia increases the risk of cardiovascular events for patients. GLP-1 (glucagon like peptide-1) is a kind of incretin discovered in recent years. It was reported that beside its hypoglycemic and losing weight effects, activator of GLP-1 receptor could decrease blood pressure and improve lipid metabolism. Sleeve gastrectomy can improve the level of blood glucose and serum lipid of type 2 diabetic rats by ameliorate insulin level and insulin resistance, which may be related with the change of gastrointestinal hormones such as ghrelin and GLP-1. So, intervention of gastrointestinal tract and gastrointestinal hormone secretion may be a new therapy for glycolipids disorder and vascular complications. But, it is lack of evidence-based medicine proof on the relationship between prokinetic drug and glycolipids metabolism. So, the investigators designed a prospective, randomized, double-blinded, placebo control study, and try to evaluate the effects of prokinetic drug (Mosapride) on the blood glucose and serum lipid in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age between 30-65 years old
* Type 2 diabetes
* Duration of diabetes less than 5 years and pancreatic function be in compensated stage.
* 7%≤HbA1C≤9%
* Patients are able to control diet and exercise by themselves in intervention period.

Exclusion Criteria:

* Type 2 diabetes with serious complications, such as diabetic neuropathy, diabetic retinopathy, stage IV diabetic nephropathy, or acute diabetic complications.
* Type 2 diabetes using insulin, GLP-1 analogues or DPP-IV inhibitors).
* Heart function in NYHA Grade II-IV or history of cardio-cerebral vascular events such as congestive heart failure, myocardial infarction or stroke within 3 months.
* Hypohepatia (AST or ALT is two times higher than the upper limit) or history of cirrhosis, hepatic encephalopathy, esophageal varices or portal shunt.
* Renal insufficiency ( serum creatinine is 1.5 times higher than the upper limit) or history of dialysis and nephritic syndrome.
* Chronic obstructive pulmonary disease (COPD), chronic respiratory failure or hyoxemia.
* Acute infections, tumor, severe arrhythmia, mental disorders, alcohol or medicine addiction.
* Fertile woman without contraceptives.
* Any surgical or medical conditions that significantly influence absorption, distribution, metabolism or excretion of the intervention drugs.
* Allergic to or have contraindication to the intervention drugs.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change of fasting plasma glucose (FPG,mmol/L) | Baseline, 24weeks (End of Trial)
Change of OGTT 2 hour blood glucose(mmol/L) | Baseline, 24weeks (End of Trial)
Change of HbA1c(%) | Baseline, 24weeks (End of Trial)
Change of control rate of blood glucose(%) | Baseline, 24weeks (End of Trial)

SECONDARY OUTCOMES:
Change of insulin release(uU/mL) | Baseline, 24weeks (End of Trial)
Change of C peptide release(nmol/L) | Baseline, 24weeks (End of Trial)
Change of HOMA-β[HOMA-β=20×（FINS,mIU/L）/（（FPG,mmol/L）-3.5）] | Baseline, 24weeks (End of Trial)
Change of HOMA-IR [HOMA-IR=(FPG,mmol/L）×（FINS,mIU/L）/22.5] | Baseline, 24weeks (End of Trial)
Change of blood glucose variability(%) | Baseline, 24weeks (End of Trial)
Change of triglyceride(mmol/L） | Baseline, 24weeks (End of Trial)
Change of total cholesterol(mmol/L） | Baseline, 24weeks (End of Trial)
Change of LDL-c(mmol/L） | Baseline, 24weeks (End of Trial)
Change of HDL-c(mmol/L） | Baseline, 24weeks (End of Trial)
Change of Glucagon(pg/ml). | Baseline, 24weeks (End of Trial)
Change of GLP(pg/ml). | Baseline, 24weeks (End of Trial)
Change of GIP(pg/ml). | Baseline, 24weeks (End of Trial)
Change of DPP-IV(pg/ml). | Baseline, 24weeks (End of Trial)
Change of waist circumference (WC,cm) | Baseline, 24weeks (End of Trial)
Change of body mass index (BMI=weight(kg)/[height(m)2], kg/m2) | Baseline, 24weeks (End of Trial)
Change of body fat(%). | Baseline, 24weeks (End of Trial)
Change of carotid intima-media thickness (IMT,mm). | Baseline, 24weeks (End of Trial)
Change of 24-hours urine sodium(mmol/24h) | Baseline, 24weeks (End of Trial)
Change of 24-hours microalbumin(mg/L). | Baseline, 24weeks (End of Trial)
Change of 24-hours mALB/Cr(mg/g.Cr). | Baseline, 24weeks (End of Trial)
Change of inflammatory markers(hs-CRP,mg/L). | Baseline, 24weeks (End of Trial)
Incidence rate of newly-diagnosed hypertension(%). | Baseline, 24weeks (End of Trial)
Heart rate variability(HRV,%). | Baseline, 24weeks (End of Trial)
Change of clinic blood pressure and 24h mean blood pressure(mmHg). | Baseline, 24weeks (End of Trial)

CONTACTS AND LOCATIONS:
Overall Officials: Zhu Zhiming, MD, PhD, Study Director — The third hospital affiliated to the Third Military Medical University. China